CLINICAL TRIAL: NCT03345238
Title: Neurophysiological Effects of Dry Needling in Patients With Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Rey Juan Carlos (Other)
Collaborators: Luis Martín Sacristán (Unknown)
Responsible Party: Principal Investigator, Josue Fernandez Carnero, Tesis Director, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 31/8/2017
Record Dates: First submitted 2017-08-31; First posted 2017-11-17 (Actual); Last update posted 2019-11-12 (Actual); Status verified 2019-11

CONDITIONS: Myofascial Pain Syndrome
Keywords: Dry Needling; Myofascial Pain Syndrome; Neurophysiological effects; Autonomic Nervous System
MeSH Terms: conditions — Myofascial Pain Syndromes

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with double-blind
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active MTP (Experimental)
  Interventions: Procedure: Deep Dry Needling
- Latent MTP (Experimental)
  Interventions: Procedure: Deep Dry Needling
- Out of MTP (Experimental)
  Interventions: Procedure: Deep Dry Needling

INTERVENTIONS:
Procedure: Deep Dry Needling — Deep Dry Needling in the upper trapezious muscle is an invasive technique of Physical Therapy.

SUMMARY:
The present study aims to evaluate the differences that may be experienced in pain and cervical disability, before, during and just after the intervention of the Deep Dry Needling in the upper trapezius muscle in active, passive myofascial trigger points (MTP) or non-MTP in Patients with neck pain, assessing, in turn, the neurophysiological effects on the Autonomic Nervous System.

Hypothesis: Deep Dry Needling of active myofascial trigger points produces a greater decrease of pain and cervical disability index and increase of pressure pain threshold; Than the Deep Dry Needling of Myofascial Trigger Points latent or out of Myofascial Trigger Points in patients with chronic neck pain.

Objective: To determine the efficacy of Deep Dry Needling applied on Active Myofascial Triggers (MTP) vs. latent MTP versus MTP, on pain reduction and cervical disability, in patients with chronic neck pain attributable to Myofascial Pain Syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Non-specific neck pain, unilateral or bilateral.
* Neck pain ≥ 3 months of duration.
* Presence of active and latent MTP in the upper, left, right or bilateral trapezius muscle, in relation to the patient's neck pain.
* Clinical criteria recommended to identify active and latent MTP:

  1. Tensile band palpable.
  2. Exquisite local pain at the pressure of a taut band node.
  3. Recognition by the patient of their usual pain when pressing on the sensitive nodule (to identify an active MTP).
  4. Painful limitation of range of mobility to complete stretching. It is considered positive when 3 of the 4 clinical criteria are found.

Exclusion Criteria:

* Unsurpassed fear of needles.
* Coagulation disorders.
* Specific alterations of the cervical region in the clinical history.
* Infiltration of corticosteroids or local anesthetics during a year before the study.
* Surgical intervention of the cervical region or previous shoulder.
* Skin lesions in the area, as well as infection or inflammation.
* Taking analgesic, anti-inflammatory or anticoagulant medication the week before the study.
* Treatment of MTP or Deep Dry Needling in the neck region in the 6 months prior to the intervention.
* Cognitive deficit in the medical history.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2017-03-13 (Actual); Primary Completion 2017-12-29 (Actual); Study Completion 2019-08-10 (Actual)

PRIMARY OUTCOMES:
Efficacy of Deep Dry Needling applied on Active Myofascial Trigger Points (MTP) vs. latent MTP versus outside MTP, on pain reduction in patients with chronic neck pain. | Baseline, during intervention, immediately after intervention, 1, 6, 12, 24, 48 and 72 hours after intervention, a week after intervention and one month after the intervention
  Checkin the Intensity of pain with the Visual Analogic Scale.
  It is a 100 mm line that measures the intensity of pain.The left end of the line represents the absence of pain, while the far right represents the worst pain imaginable. The numerical scale of intensity of pain adds a numerical ranking where 1 is no pain and 10 the worst pain imaginable.

SECONDARY OUTCOMES:
Threshold of pain to pressure | Baseline and immediately after intervention
  Using a Digital algometer in the pain points of the patient.
Cervical pain and dysfunction | Baseline, a week after intervention and one month after the intervention
  Using the questionnaire: Neck Disability Index
  It is the scale that has been used in more different populations and the one that has been more times validated against multiple measures of function, pain and clinical signs and symptoms. The NDI is a self-completed questionnaire with 10 sections. Each of the sections (cervical pain intensity, personal care, weight lifting, reading, headache, ability to concentrate, work capacity, driving, sleep and leisure activities) offers 6 possible answers that represent 6 levels progressive functional capacity, and scored from 0 to 5 (0 = no disability, 5 = total disability). The total score is expressed in percentage terms with respect to the maximum possible.
Cervical pain and dysfunction | Baseline
  Using the questionnaire: Catastrophic Scale of Pain
  It is a self-administered scale of 13 items and one of the most used to assess the construct "catastrophization in the face of pain".
  It comprises 3 dimensions: a) rumination; b) magnification, and c) hopelessness.
  The theoretical range of the instrument is between 13 and 62, indicating low scores, little catastrophization, and high values, high catastrophization.
Cervical pain and dysfunction | Baseline, a week after intervention and one month after the intervention
  Using the questionnaire: Chronic pain gradation scale
  It is a scale that serves as a valid, reliable and useful instrument to measure chronic pain early in clinical practice. The first factor formed by 4 items, can be called "disability related to pain"; the second, "the intensity of pain", is made up of 3 items. The version of the scale in Spanish consists of 8 items and the final score is obtained with the sum of items 2 to 8, which results in a range of 0 to 70.
Changes related to the Autonomic Nervous System | Baseline, during intervention and after intervention (1 and 10 minutes after intervention)
  Checking heart rate measuring the beats per minute.
Changes related to the Autonomic Nervous System | Baseline, during intervention and after intervention (1 and 10 minutes after intervention)
  Checking changes of the skin temperature measuring the surface temperature of the skin in ºC.
Changes related to the Autonomic Nervous System | Baseline, during intervention and after intervention (1 and 10 minutes after intervention)
  Checking changes on skin conductance measuring the conductance of the skin in microsiemens.

CONTACTS AND LOCATIONS:
Overall Officials: Luis Martín Sacristán, MSc, Principal Investigator — University of Alcala
Locations (1):
- universidad de Alcalá de Henares, Alcalá de Henares, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No